CLINICAL TRIAL: NCT06653465
Title: Intravenous Acetaminophen for Postoperative Delirium in Older Patients Recovering From Major Noncardiac Surgery: a Randomised Controlled Study
Brief Title: Intravenous Acetaminophen for Postoperative Delirium in Older Patients Recovering From Major Noncardiac Surgery
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LY-2023-239
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Delirium in Old Age
Keywords: postoperative delirium; acetaminophen; elderly patient
MeSH Terms: conditions — Emergence Delirium | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intravenous aceteminophen group (Experimental): 50 ml contains 500 mg of acetaminophen will be administered for the first dose when the surgical suture begin at the end of surgery and thereafter repeated every 6 hours for the following 7 doses using automatic intravenous pump (4g acetaminophen diluted with 0.9% saline to 400 ml), and every bolus of 50 ml will be finished within 10 minutes.
  Interventions: Drug: Acetaminophen
- saline placebo group (Placebo Comparator): 50 ml 0.9% saline will be administered for the first dose placebo when the surgical suture begin at the end of surgery and thereafter repeated every 6 hours for the following 7 doses using automatic intravenous pump (400ml 0.9% saline without acetaminophen), and every bolus of 50 ml will be finished within 10 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen, which has similarly effects with NSAIDs in terms of inhibition of cyclooxygenase COX1, COX2 and COX3, is widely used as adjuvant for perioperative multimodal analgesia.
  Arms: intravenous aceteminophen group
Drug: Saline — Saline, a kind of crystalloid widely used in clinical treatment.
  Arms: saline placebo group

SUMMARY:
Investigators propose this multi-center randomised controlled study to test the preventive effect of intravenouse acetaminophen in delirium over 5 postoperative days among older patients recovering from major non-cardiac surgery.

DETAILED DESCRIPTION:
Delirium is a common complication in elderly patients after major surgeries and can lead to poor outcomes such as neurocognitive decline. Acetaminophen is a widely used adjuvant for perioperative multimodal analgesia. It can effectively alleviate postoperative pain, promote opioid-sparing and exert anti-neuroinflammatory response, showing strong potential for preventing postoperative delirium. There is evidence that intravenous acetaminophen reduces delirium in older patients following cardiac surgery, but its effectiveness is inconclusive among non-cardiac surgical patients. Investigators propose this multi-center, randomized, placebo-controlled, parallel-group trial in patients aged >65 years old scheduled for non-cardiac major surgery with general anesthesia expected to last at least 2 h. A total of 1930 elderly patients will be enrolled and randomized at 1:1 ratio to acetaminophen or saline placebo groups, stratified by age, education level, and trial site with random-sized blocking. Acetaminophen or saline will be given when the surgical suture begin at the end of surgery and thereafter a total of 7 doses within 48h after surgery. The primary outcome will be the incidence of delirium, assessed twice daily, through the five postoperative days. Secondary outcomes will include pain scores with movement, opioid use within the first 48 postoperative hours, severity of delirium, ICU and hospital lengths of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years.
2. Scheduled for non-cardiac major surgery with general anesthesia that is expected to last more than 2h.
3. ASA Physical Status I-III.
4. Weight >50 kg.
5. Written informed consent.

Exclusion Criteria:

1. Pre-existing neuropsychiatric diseases (Alzheimer's disease, Schizophrenia, Parkinson's Disease, Seizures, etc.).
2. Pre-existing cognitive impairment (MMSE<18).
3. Preoperative delirium.
4. Severe circulatory instability (preoperative left ventricular ejection fraction less than 30%, unstable angina, severe coronary artery disease, sick sinus syndrome, etc.).
5. Contraindication to the acetaminophen use, including serum creatinine > 177µmol/L or aminotransferses > 3 times the upper limit of normal.
6. Alcohol or drug abuse within a year before surgery.
7. Inability to communicate because of severe visual/auditory dysfunction or language barrier.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1930 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Participants will be followed up during the first 5 postoperative days.
  Delirium will be assessed by the trained investigators twice daily, from 8-10 AM and from 5-7 PM, starting from postoperative day 1 using 3-minute Confusion Assessment Method (3D-CAM) or CAM-ICU for intubated patients. Immediately before assessing delirium, sedation or agitation was assessed using Richmond Agitation-Sedation Scale (RASS). If the patient was too deeply sedated or unarousable (RASS -4 or -5), delirium assessment was aborted and the patient was recorded as comatose.

SECONDARY OUTCOMES:
Delirium type | Participants will be followed up during the first 5 postoperative days.
  Patients with delirium were classified into three motoric subtypes. Hyperactive delirium was defined when RASS was consistently positive (+1 to +4); hypoactive delirium was defined when RASS was consistently neutral or negative (-3 to 0); and mixed delirium was defined when some RASS scores were positive (+1 to +4) and some RASS scores were neutral or negative (-3 to 0).
Delirium severity | Participants will be followed up during the first 5 postoperative days.
  Delirium rating scale 98 revised (DRS-R-98) will be used to evaluate severity of delirium. DRS-R-98 consists of 16 items, including 13 items to assess severity of delirium and 3 diagnostic items. The total severity score range from zero (best) to 39 (worst).
Pain scores | Participants will be followed up during the first 5 postoperative days.
  Pain scores will be assessed using numerical rating scale (NRS) once daily, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable".
Total opioid consumption | Participants will be followed up during the first 5 postoperative days.
  Amount of intravenous and/or oral opioid consumption for analgesia will be recorded.
Delirium duration | Participants will be followed up during the first 5 postoperative days.
  Time to onset of delirium.

OTHER OUTCOMES:
Cognitive function | Cognitive function will be evaluated on the fifth day after operation.
  Cognitive function will be evaluated with Mini-Mental State Examination (MMSE) score that ranges from zero (worst) to 30 (best).
Length of days in ICU and hospital after surgery | one month
  Length of stay in ICU and hospital after surgery will be collected from electronic medical records.
All cause mortality | one month

CONTACTS AND LOCATIONS:
Overall Officials: LIQUN YANG, MD, Principal Investigator — Anesthesiology, Renji Hospital, Shanghai Jiao Tong University, School of Medicine Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be shared in peer-reviewed academic journals. Other IPD will be made available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Zheng M, Wang B, Mao M, Wu Y, Wang Z, Yang L. Intravenous acetaminophen for postoperative delirium in older patients recovering from major non-cardiac surgery: a randomised-controlled study protocol. BMJ Open. 2025 May 15;15(5):e097079. doi: 10.1136/bmjopen-2024-097079. PMID 40379334